CLINICAL TRIAL: NCT05002491
Title: Change in Leptin as a Predictor of Satiety With High Protein Feeding
Acronym: HiProLep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan Purnell, Professor, Oregon Health and Science University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: Protocol 695
Record Dates: First submitted 2021-07-20; First posted 2021-08-12 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Dietary Exposure
Keywords: protein
MeSH Terms: interventions — Diet, High-Protein

STUDY DESIGN:
Intervention Model Description: Isocaloric feeding phase followed by ad-libitum feeding phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High protein feeding (Experimental): Two isocaloric feeding phases of 2 weeks followed by an ad-libitum feeding phase of 3 months
  Interventions: Other: High protein diet

INTERVENTIONS:
Other: High protein diet — Normal vs high protein dietary feeding

SUMMARY:
Body weight can be affected by the content of fat and carbohydrate in the diet. On average, people will lose a modest (< 5 kg) amount of weight when switched from a high fat diet to a low fat, high carbohydrate diet. Determining mechanisms whereby changing the makeup of the diet can change one's body weight will be important in understanding why body weight in the US population is trending upward recently and what health care providers can recommend to reverse this trend. Previous studies have shown that increasing the carbohydrate and lowering the fat content in the diet leads to a change in the appearance of the hormone leptin in the blood over 24 hours. Leptin is an important signal from the fat cell to the brain that leads to a reduction in appetite and weight loss. A previous study found that after keeping people's weight stable, that the greater rise in leptin over the day on a low fat-high carbohydrate diet compared to a high fat diet predicted the reduction in calories they ate over a subsequent 12 weeks when their weight was allowed to freely fluctuate. Recent studies have also provided evidence that limiting fat and increasing the amount of protein in the diet also leads to modest weight loss. It is therefore proposed to test whether low fat, high protein diets also result a change in leptin secretion, and if this change predicts a reduction in appetite when they are allowed to eat freely.

DETAILED DESCRIPTION:
The role of leptin in regulating body fat mass in humans is incompletely understood. Although complete loss of leptin signaling results in morbid obesity, there is an inconsistent association between more subtle changes in leptin levels and changes in body composition. Administration of recombinant leptin to human volunteers also results in a variable loss of fat mass. Therapeutic high carbohydrate diets generally lead to decreased caloric intake and weight loss compared with high fat diets. The mechanism of this decrease in appetite is, however, unknown. In preliminary data, the invesigators have shown that compared to high fat feeding, isocaloric high carbohydrate feeding over 2 weeks leads to increased leptin excursion during 24 hours. In addition, this change in leptin signaling predicts subsequent reduction in daily caloric intake with ad-lib high carbohydrate feeding. It has recently been reported that an increase in dietary protein also leads to modest spontaneous weight loss in ad-lib feeding subjects. The current proposal is to therefore determine whether prolonged high protein feeding leads to a sustained increase in the integrated daily leptin level and whether this increase predicts a subsequent decrease in caloric intake in human volunteers. Eligible subjects will consume a control protein diet (15%, low protein) followed by a high protein diet (30% protein) for 2 weeks each while maintaining weight stability. At the end of each 2-week feeding phase, subjects will be admitted to the inpatient GCRC for frequent sampling for insulin and leptin levels over 24 hours. Immediately following the second CRC inpatient visit, subjects will continue to consume the high protein diet ad-libitum for another 12 weeks, during which time they will be followed for changes in their caloric intake and body weight. Because of limitations in metabolic kitchen resources, if this study were to be conducted solely at OHSU, it would require recruitment and study of two groups of subjects over sequential time periods. This results in delay of acquisition of data, completion of the study, and the potential introduction of seasonal variation as a study confounder. Therefore, a two-site study is proposed utilizing the metabolic kitchen resources of OHSU and the University of Washington GCRC's jointly. Instead of two groups of subjects being recruited and studied sequentially at one site, subjects will be recruited at both sites and studied in parallel, thus allowing the completion of the protocol in half the usual amount of time and without additional study confounders.

It is hypothesized that switching human volunteers from a 15% protein diet to an isocaloric high (30%) protein diet will cause a significant increase in the area under the diurnal plasma leptin versus time curve (AUC-leptin) and the insulin versus time curve (AUC-insulin), that these increases will be sustained over 2 weeks of isocaloric high protein feeding, and that the elevation in AUC-leptin will predict the extent to which caloric intake decreases when subjects are switched from an isocaloric to an ad libitum high protein diet.

Specific Aim 1: To determine whether an isocaloric increase in dietary protein content from 15% to 30% causes a significant increase in AUC-leptin and AUC-insulin that is sustained for two weeks.

Specific Aim 2: To determine whether the increase in AUC-leptin on a 30% protein diet predicts a subsequent decrease in ad libitum caloric intake and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed written consent
* Age between 18 and 65 years
* Willingness to consume only food prepared by the CRC for 6 weeks
* Body mass index between 22 and 28 kg/m2
* Weight stable to within 2 kg for 3 months preceding study, and at lifetime maximal weight

Exclusion Criteria:

* Diabetes mellitus
* Renal disease
* Other chronic medical or psychiatric illness
* Pregnancy or female subject unwilling to use contraception
* Use of tobacco products
* Regular intense exercise (>30 minutes of aerobics, 3x / week)
* Vegetarian or extreme dietary preferences (< 20% or > 40% fat diet, > 40% protein diet)
* Use of anabolic steroids, glucocorticoids, or lipid-lowering agents
* Alcohol consumption >2 drinks / day

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2002-05-01 (Actual); Primary Completion 2003-12-31 (Actual); Study Completion 2003-12-31 (Actual)

PRIMARY OUTCOMES:
24 hour levels of leptin after isocaloric and ad-libitum feeding phases | After each 2 week isocaloric feeding phase (x2) and a 3 month ad-lib feeding phase
  Change in leptin levels measured every 30 minutes while consuming diet-assigned meals
24 hour levels of ghrelin after isocaloric and ad-libitum feeding phases | After each 2 week isocaloric feeding phase (x2) and a 3 month ad-lib feeding phase
  Change in ghrelin levels measured every 30 minutes while consuming diet-assigned meals
Body weight | Weekly during each 2 week isocaloric feeding phase (x2) and a 3 month ad-lib feeding phase
  Change in body weight

SECONDARY OUTCOMES:
Appetite scores | Daily during each 2 week isocaloric feeding phase (x2) and a 3 month ad-lib feeding phase
  Changes in self-reported visual analog scores (VAS) for hunger, fullness measured every 30 minutes while consuming diet-assigned meals
Lipid levels at each study visit | Daily during each 2 week isocaloric feeding phase (x2) and a 3 month ad-lib feeding phase
  Changes in lipid levels at the end of the trial phases involving different diet-assigned meals

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weigle DS, Breen PA, Matthys CC, Callahan HS, Meeuws KE, Burden VR, Purnell JQ. A high-protein diet induces sustained reductions in appetite, ad libitum caloric intake, and body weight despite compensatory changes in diurnal plasma leptin and ghrelin concentrations. Am J Clin Nutr. 2005 Jul;82(1):41-8. doi: 10.1093/ajcn.82.1.41. PMID 16002798
- [Background] Koren MS, Purnell JQ, Breen PA, Matthys CC, Callahan HS, Meeuws KE, Burden VR, Weigle DS. Changes in plasma amino Acid levels do not predict satiety and weight loss on diets with modified macronutrient composition. Ann Nutr Metab. 2007;51(2):182-7. doi: 10.1159/000103323. Epub 2007 May 30. PMID 17541265
- [Background] Kratz M, Weigle DS, Breen PA, Meeuws KE, Burden VR, Callahan HS, Matthys CC, Purnell JQ. Exchanging carbohydrate or protein for fat improves lipid-related cardiovascular risk profile in overweight men and women when consumed ad libitum. J Investig Med. 2010 Jun;58(5):711-9. doi: 10.231/JIM.0b013e3181da4d37. PMID 20305576
- [Background] Kremsdorf RA, Hoofnagle AN, Kratz M, Weigle DS, Callahan HS, Purnell JQ, Horgan AM, de Boer IH, Kestenbaum BR. Effects of a high-protein diet on regulation of phosphorus homeostasis. J Clin Endocrinol Metab. 2013 Mar;98(3):1207-13. doi: 10.1210/jc.2012-2910. Epub 2013 Feb 7. PMID 23393178
- [Derived] Horgan AM, Palmbach GR, Jordan JM, Callahan HS, Meeuws KE, Weigle DS, Kratz M, Purnell JQ. Self-selected meal composition alters the relationship between same-day caloric intake and appetite scores in humans during a long-term ad-libitum feeding study. Eur J Nutr. 2023 Mar;62(2):1003-1009. doi: 10.1007/s00394-022-03040-5. Epub 2022 Nov 8. PMID 36346472